CLINICAL TRIAL: NCT03841708
Title: Impact on Lactate Clearance of Early Hemodynamic Optimization Through Pleth Variability Index in the ED for Resuscitated Out-of-hospital Cardiac Arrests
Brief Title: Hemodynamic Optimization Through Pleth Variability Index for OHCA
Acronym: HemOpt-PVI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stefano Malinverni, MD (Other)
Collaborators: Andre Vesale Association (Unknown)
Responsible Party: Sponsor-Investigator, Stefano Malinverni, MD, Consultant Academic Doctor, Centre Hospitalier Universitaire Saint Pierre
Organization: Centre Hospitalier Universitaire Saint Pierre (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HemOpt-PVI
Record Dates: First submitted 2019-01-30; First posted 2019-02-15 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-11

CONDITIONS: Cardiac Arrest With Successful Resuscitation
Keywords: Cardiac arrest; Hemodynamic monitoring; Non invasive monitoring; Pleth Variability Index; Adult cardiac arrest
MeSH Terms: conditions — Heart Arrest

STUDY DESIGN:
Intervention Model Description: In this monocentric placebo controlled single blind ranomized clinical trial patients will be recruited from the Emergency Department of a University Hospital.
  80 patients suffering form a out of hospital cardiac attest arriving at the Emergency Department with a lactate level > 4 mmol/L or a mean arterial pressure below 65 mmHg will be included in the study at the moment of admission to the Emergency Department and patients in the treatment arm will be monitored on top of standard monitoring with a non invasive device measuring continuously the pleth variability index(PVI). Patients in the treatment arm will be treated according to an algorithm integrating both standard non invasive measures and the PVI. Patients in the control arm will be treated according to non invasive measures only.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Pleth Variability Index (Active Comparator): In the experimental group patients will be hemodynamically resuscitated in the early phases after ROSC based on the pleth variability index on top of standard non invasive monitoring
  Interventions: Device: Pleth variability index
- Standard non invasive monitoring (Placebo Comparator): In the control group patients will be hemodynamically resuscitated in the early phases after ROSC based on standard non invasive monitoring such as SatO2, EtCO2, non invasive blood pressure and continuous ECG.
  Interventions: Device: Standard non invasive monitoring

INTERVENTIONS:
Device: Pleth variability index — The utility of a early goal directed therapy will be evaluate by the pleth variability index (PVI). If above>13% in a well sedated patients perfectly synchronized with the ventilator providing at least 6ml/kg of ideal body weight, a fluid challeng with 10ml/kg of NaCl 0,9% will be administrated. Patient will be constantly re-assessed until the hemodynamic goals of a mean arterial pressure above 65 mmHg, a capillary refill time below 3 seconds, a decreasing trend on lactates and a urinary output above 0.5/ml/kg/h will be achieved. The second fluid challenge will always be performed with 100 ml of albumin 20%. The third fluid challenge if necessary will be performed with 10 ml/kg of NaCl 0.9%.
  Other Names: Pleth Variability Index and standard non invasive monitoring
  Arms: Pleth Variability Index
Device: Standard non invasive monitoring — In the control group patients will be hemodynamically resuscitated in the early phases after ROSC based on standard non invasive monitoring such as SatO2, EtCO2, non invasive blood pressure and continuous ECG. If deemed necessary by the treating physician a fluid challenge of 10ml/kg of NaCl 0,9% will be administrated. Patient will be constantly re-assessed until the hemodynamic goals of a mean arterial pressure above 65 mmHg, a capillary refill time below 3 seconds, a decreasing trend on lactates and a urinary output above 0.5/ml/kg/h will be achieved. The second fluid challenge will always be performed with 100 ml of albumin 20%. The third fluid challenge if necessary will be performed with 10 ml/kg of NaCl 0.9%.
  Arms: Standard non invasive monitoring

SUMMARY:
Less than half of the patients suffering from sudden cardiac arrest arrive at the hospital alive. Within these survivors less than half will be discharged alive from the hospital without being severely disabled.

The most frequent cause of death during the first 24 hours since admission to the hospital is related to cardiovascular instability and failure. In the early phases of ROSC patients are hemodynamically unstable and management for out of hospital cardiac arrests relies on few non invasive measurements such as non invasive blood pressure, SatO2, EtCO2 and continuous ECG. Recent technological advances allow continuous non invasive evaluation of response to fluid challenge in mechanically ventilated patients through the pleth variability index.

The investigators hypothesize that early goal directed therapy based on non invasive measurement of the pleth variability index on top of conventional non-invasive monitor during the initial care in the Emergency Department can improve the hemodynamic status of the participants, increase lactate clearance and reduce fluid balance at 48 hours post arrest.

Objectives:

* To determine whether an early goal directed management based on the pleth variability index on top of standard non invasive hemodynamic monitoring could improve the hemodynamic status of patients post cardiac arrest especially in terms of increase in lactate clearance and reduced fluid balance. Neurological outcome will be investigated.

DETAILED DESCRIPTION:
Less than half of the patients suffering from sudden cardiac arrest arrive at the hospital alive. Of these survivors less than half will be discharged alive from the hospital without being severely disabled.

The most frequent cause of death during the first 24 hours since admission to the hospital is related to cardiovascular instability and failure. In the early phases of ROSC from out of hospital cardiac arrest patients are hemodynamically unstable and management relies on few non invasive measurements such as non invasive blood pressure, SatO2, EtCO2 and continuous ECG.

Even at arrival at the ER patients are monitored by non-invasive parameters during the early phases and invasive hemodynamic monitoring may be delayed until ICU admission. Recent technological advances allow continuous non invasive evaluation of response to fluid challenge in mechanically ventilated patients through the pleth variability index.

The research proposal by the investigator is a randomized prospective interventional, single-center study based at Saint Pierre University Hospital, carried out in the emergency department.

Participant will be OHCA admitted alive to the Emergency department with unstable hemodynamics defined as a mean systolic pressure below 70 mmHg or a blood lactate concentration of at least 36 mg/dL (4 mmol/L).

The criteria for exclusion from the study will be pregnancy, being a prisoner or having limitations of therapeutic effort.

During the study the investigators will evaluate whether an hemodynamic protocol based on pleth variability index on top of routine non invasive monitoring is superior to the routine non invasive monitoring only ( such as non invasive blood pressure, EtCO2, SatO2 and ECG) in terms of lactate clearance and fluid balance.

In both study arms the treating clinician will be encouraged to achieve and maintain the following hemodynamics goals: a mean arterial pressure above 70mmHg, a diuresis above 0.5 ml/kg/h, a capillary refill time below 3 and a clearance of lactate above 10% after 2 hours.

In the control arm the participants will be initially resuscitated with an initial bolus of NaCl 0.9% 10ml/kg whenever the patient is not meeting the set hemodynamic goals. If deemed necessary a second fluid challenge of 100 ml of Albumin 20% will be administered to the patient. Any further fluid challenge will be done with NaCl 0.9% 10ml/kg. At any moment the treating clinician will be allowed to initiate a continuous infusion of noradrenaline or dobutamine to achieve the hemodynamic goals. If deemed necessary clinicians will be allowed to perform a cardiac echography at any moment to assess the hemodynamic needs of the patient. Patients will be continuously reassessed to verify that the hemodynamic goals are achieved.

In the intervention arm patient will be resuscitated according to their PVI. Whenever the PVI will be above 13% the patient will be considered as being fluid responsive and a fluid challenge will be performed whenever the patient is not meeting the set hemodynamic goals. First fluid challenge will be an initial bolus of NaCl 0.9% 10ml/kg. If deemed necessary a second fluid challenge of 100 ml of Albumin 20% will be administered to the patient. Any further fluid challenge will be done with NaCl 0.9% 10ml/kg. If the hemodynamic goals are not achieved and the PVI is below 13% an infusion of noradrenaline will be initiated aiming at a mean arterial pressure of at least 70 mmHg. Infusion of dobutamine to achieve the hemodynamic goals will be started according to clinician decision. If deemed necessary clinicians will be allowed to perform a cardiac echography at any moment to assess the hemodynamic needs of the patient.

Patients will be continuously reassessed to verify that the hemodynamic goals are achieved.

In both arms participants will be sedated according to our hospital protocol for OHCA which includes propofol and remifentanyl titrated to achieve a good synchronization between the patient and the ventilator. If despite sedation a good synchronization between the patient and the ventilator cannot be achieved participants will be initially curarized.

Intervention will end at ICU admission when hemodynamic therapeutic decisions will be based on invasive hemodynamic monitoring.

Trainings will be organized for nurses and postgraduate doctors during the months preceding the study to familiarize the medical-nursing team with the study.

ELIGIBILITY:
Inclusion Criteria:

* Out of Hospital Cardiac Arrest
* ROSC before Emergency department admission
* Mecanically ventilated with a tidal volume of at least 6 ml/IBW
* Admitted to the emergency department with a lactate > 4mmol/L or a mean arterial pressure below 65 mmHg or a TRC>5 seconds

Exclusion Criteria:

* Minor
* Prisoners
* Pregnant woman
* Atrial fibrillation

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2023-09-01 (Actual); Study Completion 2023-09-30 (Actual)

PRIMARY OUTCOMES:
Change of lactate | From ED admission until 6 hours from admission with 1 predefined time point at 3 hours from ED admission
  Change of lactate at 3h from admission. Lactate clearance will be measured as {(Admission lactate [mmol/L] - Lactate at time point [mmol/L]) / (Admission lactate [mmol/L])} x 100

SECONDARY OUTCOMES:
Mortality 24h | 24 hours
  Mortality at 24 hours: measured as the rate of mortality during the first 24 hours from ER admission within the two study groups
Mortality 72h | 72 hours
  Mortality at 72 hour:s measured as the rate of mortality during the first 72hours from ER admission within the two study groups
Change of lactate | From ED admission until 24 hours from admission with 3 predefined time points at 6,12 and 24 hours from ED admission
  Change of lactate at 6h 12h and 24h from admission. Lactate clearance will be measured as {(Admission lactate [mmol/L] - Lactate at time point [mmol/L]) / (Admission lactate [mmol/L])} x 100. Patients dying during the observation period will be imputated a lactate clearance of 0
Fluid balance first 48 hours | 48 hours
  Fluid balance at 48 hours post ROSC. Fluid balance will be measured from treatment chart as follows: [total fluid intake from ER admission to 48 hours post ER admission (crystalloids, colloids, drugs dilution fluids) - total urine output from ER admission until 48th hours since ER admission]
Fluid balance first 24 hours | 24 hours
  Fluid balance at 24 hours post ROSC. Fluid balance will be measured from treatment chart as follows: [total fluid intake from ER admission to 24 hours post ER admission (crystalloids, colloids, drugs dilution fluids) - total urine output from ER admission until 24th hours since ER admission]
SOFA 24 hours | 24 hours
  SOFA at 24 hours post-ROSC: The Sequential Organ Failure Assessment score (SOFA) regroups six different scores one each for the respiratory, cardiovascular, hepatic, coagulation, renal and neurological systems. It ranges from 0 to 24. Higher values of the score are associated with worse outcome. It will be calculated based on laboratory and clinical values collected closest to the 24th hour since ER admission within the time window going from 18 hours to 30 hours. Since the investigators expect all patients included in this study to be intubated and sedated, GCS would be of limited value and therefore the final CPC score minus 1 will be used as the neurologic failure component.
CPC at hospital discharge | At 16 weeks or at hospital discharge whichever comes first
  CPC at hospital discharge: Cerebral Performance Category (CPC) ranges from 1 to 5. It will be recovered from hospital records describing the clinical condition at the precise moment of patient discharge. Good clinical outcome will be defined as Cerebral performance category 1 or 2 at hospital discharge.
Normalization of lactate | 48 hours
  Time measured in hours it takes from admission to reach a lactate level < 2mmol/L

CONTACTS AND LOCATIONS:
Overall Officials: Stefano Malinverni, MD, Principal Investigator — Centre Hospitalier Universitaire Saint Pierre
Locations (1):
- CHU Saint Pierre, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: Yes
The full database of the study will be accessible from the public after termination and publication of the study
Supporting Information: Study Protocol, ICF
Time Frame: Data will become available at study pubblication
Access Criteria: Open access

REFERENCES:
- [Background] Nolan JP, Soar J, Cariou A, Cronberg T, Moulaert VR, Deakin CD, Bottiger BW, Friberg H, Sunde K, Sandroni C. European Resuscitation Council and European Society of Intensive Care Medicine Guidelines for Post-resuscitation Care 2015: Section 5 of the European Resuscitation Council Guidelines for Resuscitation 2015. Resuscitation. 2015 Oct;95:202-22. doi: 10.1016/j.resuscitation.2015.07.018. No abstract available. PMID 26477702
- [Background] Gaieski DF, Band RA, Abella BS, Neumar RW, Fuchs BD, Kolansky DM, Merchant RM, Carr BG, Becker LB, Maguire C, Klair A, Hylton J, Goyal M. Early goal-directed hemodynamic optimization combined with therapeutic hypothermia in comatose survivors of out-of-hospital cardiac arrest. Resuscitation. 2009 Apr;80(4):418-24. doi: 10.1016/j.resuscitation.2008.12.015. Epub 2009 Feb 12. PMID 19217200
- [Background] Cannesson M, Delannoy B, Morand A, Rosamel P, Attof Y, Bastien O, Lehot JJ. Does the Pleth variability index indicate the respiratory-induced variation in the plethysmogram and arterial pressure waveforms? Anesth Analg. 2008 Apr;106(4):1189-94, table of contents. doi: 10.1213/ane.0b013e318167ab1f. PMID 18349191
- [Background] Rivers E, Nguyen B, Havstad S, Ressler J, Muzzin A, Knoblich B, Peterson E, Tomlanovich M; Early Goal-Directed Therapy Collaborative Group. Early goal-directed therapy in the treatment of severe sepsis and septic shock. N Engl J Med. 2001 Nov 8;345(19):1368-77. doi: 10.1056/NEJMoa010307. PMID 11794169
- [Background] Aya HD, Cecconi M, Hamilton M, Rhodes A. Goal-directed therapy in cardiac surgery: a systematic review and meta-analysis. Br J Anaesth. 2013 Apr;110(4):510-7. doi: 10.1093/bja/aet020. Epub 2013 Feb 27. PMID 23447502
- [Background] Benes J, Giglio M, Brienza N, Michard F. The effects of goal-directed fluid therapy based on dynamic parameters on post-surgical outcome: a meta-analysis of randomized controlled trials. Crit Care. 2014 Oct 28;18(5):584. doi: 10.1186/s13054-014-0584-z. PMID 25348900
- [Background] Yin JY, Ho KM. Use of plethysmographic variability index derived from the Massimo((R)) pulse oximeter to predict fluid or preload responsiveness: a systematic review and meta-analysis. Anaesthesia. 2012 Jul;67(7):777-83. doi: 10.1111/j.1365-2044.2012.07117.x. Epub 2012 Mar 27. PMID 22452345
- [Result] Topjian AA, Berg RA, Taccone FS. Haemodynamic and ventilator management in patients following cardiac arrest. Curr Opin Crit Care. 2015 Jun;21(3):195-201. doi: 10.1097/MCC.0000000000000205. PMID 25887300
- [Result] Loupec T, Nanadoumgar H, Frasca D, Petitpas F, Laksiri L, Baudouin D, Debaene B, Dahyot-Fizelier C, Mimoz O. Pleth variability index predicts fluid responsiveness in critically ill patients. Crit Care Med. 2011 Feb;39(2):294-9. doi: 10.1097/CCM.0b013e3181ffde1c. PMID 21057311
- [Result] Zimmermann M, Feibicke T, Keyl C, Prasser C, Moritz S, Graf BM, Wiesenack C. Accuracy of stroke volume variation compared with pleth variability index to predict fluid responsiveness in mechanically ventilated patients undergoing major surgery. Eur J Anaesthesiol. 2010 Jun;27(6):555-61. doi: 10.1097/EJA.0b013e328335fbd1. PMID 20035228
- [Derived] Malinverni S, Dumay P, Domont P, Claus M, Herpain A, Grignard J, Matta S, Bouazza FZ, Ochogavia Q. Postresuscitation pleth variability index-guided hemodynamic management of out-of-hospital cardiac arrest survivors: A randomised controlled trial. Resusc Plus. 2025 Mar 19;23:100933. doi: 10.1016/j.resplu.2025.100933. eCollection 2025 May. PMID 40230365